CLINICAL TRIAL: NCT02308917
Title: The Canadian Children Inflammatory Bowel Disease Network (CIDsCaNN): A Partnership With the CH.I.L.D. Foundation: Multi-center Inception Cohort Study
Brief Title: The Canadian Children Inflammatory Bowel Disease Network (CIDsCaNN)
Acronym: CIDsCaNN
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); British Columbia Children's Hospital (Other); Alberta Children's Hospital (Other); Stollery Children's Hospital (Other); IWK Health Centre (Other); Montreal Children's Hospital of the MUHC (Other); St. Justine's Hospital (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); Eastern Health (Other); Children's Hospital of Western Ontario (Other); McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Anne Griffiths, Division Head, Gastroenterology, Hepathology and Nutrition, The Hospital for Sick Children
Other Study IDs: 1000039604
Record Dates: First submitted 2013-10-29; First posted 2014-12-05 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn's; Ulcerative Colitis
Keywords: IBD-U; Crohn's; Ulcerative colitis; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 144 Months
Biospecimen Retention: Samples With DNA — Blood samples Stool samples Biopsy Samples Colonoscopy Washing Samples Colonoscopy Brushing Samples Resection Tissue Urine Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CIDsCaNN Network is being established with the major goals of identifying why IBD develops so commonly in children and adolescents living in Canada, and of determining the best treatment strategies for different types of IBD. Focusing on a prospective, inception cohort of Canadian children of widely varied racial origins provides a unique opportunity to explore environmental risk factors early in life and close in time to disease onset, their influence on the host microbiome, and in the context of genetic susceptibility. In keeping with current treatment targets, assessed outcomes will include not only symptom resolution and growth, but also intestinal healing. We aim to identify best practice and to institute processes for continual improvement in care nationally.

DETAILED DESCRIPTION:
IBD is also known as Crohn's Disease or Ulcerative Colitis. Please read the definitions of each of these conditions below:

1. Crohn's Disease: A condition that causes "inflammation" which is swelling, redness, soreness, in different parts of your intestines; either the large intestine only, the small intestine only or both.
2. Ulcerative Colitis: A condition that causes "inflammation" which is swelling, redness and soreness in the lining of your large intestine (colon) only.

IBD may run in families, meaning that it can be passed down through genes. However, compared to other parts of the world, it has been found that the number of children with IBD living in Canada is higher. It has also been found that children whose families have come from parts of the world where IBD is not common, have the same chance of developing IBD as children born and raised in Canada. This seems particularly true for children, whose families have come here from South Asia. Because of this, doctors think that aside from genetic factors, there may be factors in the environment to explain why this has been observed.

At this time, the factors in the environment which can trigger the development of IBD are not well understood. By working together in the Network, physicians who treat IBD will be able to gain a better understanding of the environmental factors that contribute to the development of IBD.

We aim to enroll children and teenagers who have developed IBD and are being treated at participating Network centers in Canada with the goal of sharing biological samples, demographic and lifestyle information, disease history, and treatment outcomes.

Samples may be stored indefinitely so that, as additional genes, biomarkers, and microbes are discovered, their role in intestinal disease can be assessed. The importance of these samples increase over time as outcomes of intestinal disease and treatment may be tracked. As required in future, research studies proposing to use biobank data and/or samples will be submitted to a study committee and the REB (Research Ethics Board) for approval.

Approximately 2400 participants will be recruited to the Networks Inception Cohort study. They will be followed from recruitment until transfer to adult care.

The National Coordinating Centre Team and Organizational Structure

The Network's National Coordinating Centre is housed at The Hospital for Sick Children, University of Toronto. Information Technology infrastructure and support will be provided by the SickKids Research Institute's Research IT Department. Additional 'ad-hoc' resources related to IT development/support, legal counsel, bio-statistical assistance will be available to the centre as required via the resources of the SickKids Research Institute.

The National Coordinating Centre is responsible for data-integrity and completeness and ensures accountability by sites for full and timely data completeness. Support systems for collecting and recording data and encourages 'real-time' data abstraction and direct data entry. The Network is utilizing the REDCap (Research Electronic Data Capture) application as its primary data-collection platform. REDCap is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data download to common statistical packages; and 4) procedures for importing data from external sources. Within the data collection platform, numerous 'real-time' and 'post hoc' data check procedures will be implemented. Statistics concerning 'data-integrity' will be reported to the Executive Committee on a regular and frequent basis. The National Coordinating Centre will conduct site-specific staff training at the initiation of the study, when new staff are employed, and when any new tools or significant study procedures are added to the protocol.

ORGANIZATION and GOVERNANCE of NETWORK

Preamble: During the next 5-year period, the Network Executive will aim to provide both the opportunity and governance to foster development of new leaders in pediatric IBD in Canada; continue to lead in pediatric IBD research; and initiate a plan for sustainability in leadership and research productivity/funding. Diversity in the broadest sense, inclusiveness and engagement will be core values for performance. Taken together, the proposed Network governance has been changed in the following ways:

1. A plan for regular renewal of the 3-person Executive committee, which going forward will always consist of 2 co-chairs and a co-chair elect.
2. A Steering Committee (composed of committee leads or co-leads and with two additional early career representatives) will be formed in which each committee will be responsible for specific academic areas and will develop a process for renewal of its leadership. The Steering Committee will meet on a monthly basis and report to the Executive committee to update progress in their areas of responsibility and the two bodies together will drive Network activities and plans.
3. A more comprehensive, broader-ranging committee structure with clear responsibilities and deliverables.

1) 3-person Executive committee The 3-person executive committee is responsible for the overall directions, operation, and decisions of the Network. In a Network that aims to be sustainable, it is mandatory that there be a mechanism for renewal and revitalization of such leadership.

For the sake of continuity, heading into phase 2, the previous Chair (Griffiths) and one Co-chair (Mack) of the former Network Management Committee (NMC) will remain on the Executive Committee as Co-chairs. A nomination committee, consisting of Drs. David Mack, Anthony Otley, and Sally Lawrence, geographically representing respectively Central, Eastern and Western Canada, will establish a slate of candidates for the Co-chair elect position to be voted on by the Network membership in the context of the late fall annual meeting. Process for voting to be established at late August steering committee meeting.

In general, as the Network continues in the future, an elected incoming Co-chair elect, will serve on the Executive committee for 3 years (one year as co-chair Elect; two years as Co-chair), long enough to allow success in leadership, but short enough so that the opportunity for such leadership is open to the many qualified individuals within the Network, which will enrich the reach and impact of the Network efforts. As a new Chair-elect joins the 3-person executive committee, the longest serving Co-chair moves off, having in general served for 3 years.

The first co-chair Elect will join Drs Griffiths and Mack on the Executive committee in the late fall of 2021. Given the crucial period of the upcoming two years, this Executive committee will exceptionally remain in place until fall of 2023 (rather than 2022, as would happen in general). The delayed movement of Dr. Griffiths off the Executive committee and correspondingly delayed second election of a new member will mean that the 2021 co-chair elect will exceptionally serve in leadership for 4 years instead of the customary three years.

2) Steering committee Members of the Steering Committee are either committee Leads or (for larger committees) Co-Leads, with the exception that two positions are reserved for early career representatives (one representing Basic Research; one representing Clinical and Translational research). These are all named in Figure. The early career representatives, chosen based on their abilities, accomplishments and contributions to the Network to date, are affiliated with committees, but are not being given administrative responsibilities for committee leadership. It is anticipated that they will contribute meaningfully to Steering committee discussions in these roles, which have been developed as part of the Network's commitment to Training and Mentoring of the next generation of leaders.

At monthly joint meetings of the Steering and Executive committees, the expectations are 1) that committee leads will report on their activities and 2) all members together will discuss and make decisions about Network initiatives.

This change in governance structure is being made for four main reasons: 1) to allow more regular and more productive interactions between leaders with clinical investigative expertise and those with basic research expertise, given the phase 2 mandate to ensure optimal utilization of collected biospecimens, 2) to allow delegation of responsibilities with accountability, thereby aiming to increase transparency and productivity 3) to allow for greater engagement of Canadian pediatric IBD sub-specialists to find solutions for pediatric IBD, to further standardize care and 4) to foster development of new and emerging leaders.

3) Broader committee structure As shown in the Figure, the scope of committee involvement has increased from the time of Network initiation to now include Clinical care and research; Education; Patient engagement and advocacy; Training and Mentorship in addition to the prior (but somewhat renamed and refocused) Basic and Translational Research; Data management and integration; Health services research. Committees with larger portfolios will have co-leads, with shared responsibilities.

Basic and Translational research committee (BTRC): Co-Leads: Bruce Vallance and Eytan Wine Clinical care and research committee (CCRC): Co-leads, Hien Huynh and Wael El-Matary Data Management and Integration: Lead,: Thomas Walters Health Services Research: Lead, Eric Benchimol Training and Mentorship: Lead, Kevan Jacobson Education: Co-leads, Colette Deslandres and Sally Lawrence Patient engagement and advocacy: Lead, Anthony Otley

The Network remains primarily a Network for research aimed at enhancing clinical outcomes, be it development of disease prevention strategies or superior treatment paradigms. It is committed to encouraging individuals to drive specific questions using the infrastructure provided and drawing on a larger patient base than is available in individual centres. A robust data management platform with feedback of data to sites will support collection and utilization of biospecimens for basic research. Consent for linkage of data/samples to administrative health data will facilitate long-term follow-up.

An important improvement in Governance structure is the planned crosstalk between committees (e.g., ensuring mutual input between BTRC and CCRC projects), which will be achieved through the steering committee meetings as well as via co-membership in lead committees.

The addition of network-wide virtual educational initiatives over the past year has demonstrated that this is an effective way of engaging more physicians, researchers, and allied healthcare professionals in the Network. We anticipate that such interactive educational sessions will in turn 1) encourage greater engagement in prospective research and 2) provide a forum wherein data generated within the Network's studies will be shared, thereby stimulating further research and benefiting the clinical care of other patients nationally.

We anticipate that the Patient engagement and advocacy committee will have similar impact within the network.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with IBD - Crohn's, ulcerative colitis or inflammatory bowel disease undefined

Exclusion Criteria:

* Refusal to give informed consent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The network will enroll all children and adolescents diagnosed with IBD - Crohn's, Ulcerative Colitis or inflammatory bowel disease undefined (Paris A1a or A1b definitions of age at diagnosis) at participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Sustained Clinical Remission | 18 months after enrollment onto study
  Primary outcome: To test the research hypothesis, the primary endpoint is sustained clinical remission, as defined for CD by PCDAI <10 and for UC as PUCAI < 10 at each of the 6, 12, and 18 month visits AND physician global assessment of interval disease severity as quiescent at each of these visits. This primary endpoint will be assessed at 18 months, although it is the intent of the network to continue evaluations of the cohort until transfer to adult care.

SECONDARY OUTCOMES:
Other Clinical Outcomes (combination of Pediatric Crohn's Disease Activity Index, Pediatric Ulcerative Colitis Activity Index, physician global assessment of disease activity, serologic inflammatory markers and fecal calprotectin results) | 18 months after initial enrollment onto study
  Initial treatment response will be assessed at 30 days using a combination of PCDAI (Pediatric Crohn's Disease Activity Index), PUCAI (Pediatric Ulcerative Colitis Activity Index), physician global assessment of disease activity, serologic inflammatory markers and fecal calprotectin results where applicable. Information from ongoing studies shows that 60% of patients are in a sustained clinical remission by 12 months. These results will identify the percentage of patients at achieve initial treatment response within 30 days.

OTHER OUTCOMES:
Assessment of Intestinal Healing | 18 months after initial enrollment onto study
  Assessment of intestinal healing will be captured at Network Sites. Sites will be asked annually to record whether or not reassessment via endoscopy and/or MR imaging have/ has been performed and, if so, to record findings using the multi-item measures as at time of diagnosis. After 4 years of study initiation, the results will be analysed to ascertain whether including assessment using endoscopy and/or MR imaging is more accurate than assessing clinical symptoms and signs alone.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Griffiths, MD, FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (12):
- Canada (12):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Stollery Children'S Hospital, Edmonton, Alberta
  - Children'S Hospital of Bc, Vancouver, British Columbia
  - Winnipeg Children'S Hospital, Winnipeg, Manitoba
  - Janeway Children'S Health & Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - Izaak Walton Killam Hospital (Iwk), Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - CHILDRENS HOSPITAL OF WESTERN ONTARIO, Lawson Health Research Institute, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - SickKids Hospital, Toronto, Ontario
  - Montreal Children'S Hospital, Montreal, Quebec
  - Hopital Ste. Justine, Montreal, Quebec